CLINICAL TRIAL: NCT02717026
Title: Retinal Vessel Morphology in Multimodal Imaging
Brief Title: Multimodal Imaging of Retinal Vessels
Acronym: MIR
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 27-262ex14/15
Record Dates: First submitted 2015-09-07; First posted 2016-03-23 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Retinal Blood Vessels; Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Tomography, Optical Coherence; Fluorescein Angiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Optical coherence tomography — Sections including the retinal vasculature will be taken.
Device: Fluorescein angiography — Video fluorescein angiography from one eye of each subject will be performed
Device: Fundus photography — 30 and 50 degree fundus images

SUMMARY:
Retinal blood flow measurement is of scientific and clinical value. For this purpose retinal vessel morphology (such as diameter, vessel wall thickness, etc) determination is crucial. Different imaging modalities might provide divergent results. Thus, quantification of such differences is valuable.

The present study aims to reveal and quantify differences in vessel morphology between fundus photography, fundus angiography, and optical coherence tomography in health and disease.

DETAILED DESCRIPTION:
This is considered a pilot study and will pe performed on patients scheduled for routine fluorescein angiography.

During the study day the following procedures will be performed:

* Medical history and concomitant medication
* Blood pressure and heart rate
* Assessment of visual acuity using Snellen vision charts
* Biomicroscopy
* Intraocular pressure
* Funduscopy
* IOL-Master axial length measurement
* Fundusphotography
* Optical coherence tomography
* Fluorescein Angiography Fundus photography analysis will be performed with an automated software and analysis of both angiography and optical coherence tomography will be performed via the devices inbuilt software.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent, clear media

Exclusion Criteria:

* any abnormality preventing reliable vessel measurement, pregnancy,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients scheduled for routine retinal assessment
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
retinal vessel diameter | 5 minutes

SECONDARY OUTCOMES:
retinal vessel reflectivity | 5 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No